CLINICAL TRIAL: NCT00145418
Title: Phase 2 Study Evaluating the Safety and Efficacy of Eloxatin (Oxaliplatin) and Docetaxel as First-line Therapy of Stage IV or IIIB Unresectable Non-Small Cell Lung Cancer
Brief Title: Oxaliplatin and Docetaxel as First-line Therapy for Advanced Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Oncology Specialists, S.C. (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Principal Investigator, Oncology Specialists, S.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX-03-137 (0409); NCT00393081 (obsolete NCT alias)
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non small Cell Lung Cancer Stage IIIb and IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Oxaliplatin + Docetaxel as first line therapy of Stage IV or IIIB unresectable non-small cell lung cancer. The primary objective of the trial is to determine the response rate by RECIST criteria to the combination of oxaliplatin and docetaxel in patients with previously untreated NSCLC.
  Interventions: Drug: Oxaliplatin + Docetaxel

INTERVENTIONS:
Drug: Oxaliplatin + Docetaxel — Oxaliplatin 85mg/m2 Docetaxel 30mg.m2
  Other Names: Eloxatin

SUMMARY:
It has been accepted and proven that patients with unresectable lung cancer can benefit from systemic chemotherapy. Traditional platinum-based therapy has significant side effects. Oxaliplatin and docetaxel have both shown to be effective for lung cancer. The purpose of this study is to determine if oxaliplatin combined with docetaxel has a lower toxicity profile and to determine the response rate to this study drug combination.

DETAILED DESCRIPTION:
This study is a Phase II study designed to evaluate the toxicity profile for oxaliplatin and docetaxel and to determine the response rate to this study drug combination. The primary objective of the study is response rate by RECIST criteria. The secondary objective is time to progression, duration of response, and toxicity. Patients will receive:

* oxaliplatin 85mg/m2 over 2 hours on Days 1 and 15
* docetaxel 30mg/m2 on Days 1 and 8

Cycles are to be repeated every 28 days for a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small-cell lung cancer (NSCLC)
* Patients must have measurable disease
* Age greater than or equal to 18 years
* ECOG performance score of 0, 1, or 2
* Absolute neutrophil count (ANC) > 1,500
* Platelets > 100,000
* Serum creatinine < 1.5mg/dL
* Serum total bilirubin < 1.5mg/dL
* Alkaline phosphatase < 3 times the upper limit of normal
* SGOT/SGPT < 3 times the upper limit of normal
* Patients must be recovered from the effects of any prior surgery or RT.
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.
* Patients of childbearing potential and their partners must agree to use an effective form of contraception during the study and for 90 days following the last dose of study medications.

Exclusion Criteria:

* Patients with an active infection > 38.5 degrees Celsius within 3 days of the first scheduled day of protocol treatment
* Patients with active central nervous system (CNS) metastasis. Patients with stable CNS disease, who have undergone radiotherapy at least 4 weeks prior to the planned first protocol treatment and who have been on a stable dose of corticosteroids for 2 weeks are eligible for the trial.
* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin; cervical intra-epithelial neoplasm, or localized prostate cancer with a current prostate specific antigen (PSA) of < 1.0 mg/dL
* Patients with known hypersensitivity to any of the components of oxaliplatin or docetaxel
* Patients who have had prior chemotherapy for lung cancer
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment
* Grade 2 peripheral neuropathy
* Patients who are pregnant or lactating
* Any other medical condition, including mental illness or substance abuse deemed by the investigator to be likely to interfere with the patients' ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results
* History of allogeneic transplant
* Known HIV, hepatitis B or C (active, previously treated, or both)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-02; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, SC
Locations (1):
- Oncology Specialists, SC, Park Ridge, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients recruited from clinical practice.
Pre-assignment Details: patients were screened to see if they met eligibility criteria. If criteria met, enrolled into study. Otherwise listed as screen failures.
Groups:
- Oxaliplatin + Docetaxel: Oxaliplatin + Docetaxel as first line therapy of Stage IV or IIIB unresectable non-small cell lung cancer. Oxaliplatin:85 mg/m2 on Days 1 and 15 every 28 days Docetaxel:30 mg/m2 on Days 1 and 8 every 28 days.Doses will be calculated using actual body weight unless in the investigators opinion it would be in the patient's best interest to use ideal body weight. Cycles will be repeated every 28 days for a maximum of 6 cycles.
Period: Overall Study
Arm/Group | Oxaliplatin + Docetaxel
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Oxaliplatin + Docetaxel: Oxaliplatin + Docetaxel as first line therapy of Stage IV or IIIB unresectable non-small cell lung cancer
Arm/Group | Oxaliplatin + Docetaxel
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate by RECIST criteria to the combination of oxaliplatin and docetaxel in patients with previously untreated NSCLC. Per RECIST 1.0 defines a complete response (CR)as the disappearance of all disease. A partial response(PR) as a minimum of a 30% decrease in the sum of the longest dimension of target lesions. Progressive disease (PR) is defined as a minimum of a 20% increase in the sum of the longest dimension of target lesions. Stable disease is defined as neither sufficient shrinkage to qualify as a PR nor sufficient increase to qualify as PD.
Time Frame: Response is measured every 2 cycles until disease progression
Measure: Number; unit: Participants
Arm/Group | Oxaliplatin + Docetaxel
Number analyzed (Participants) | 15
Participants
  partial response | 7
  complete response | 0
  stable disease | 1

2. Secondary Outcome: Time to Progression
Description: Progression is measured from each participants start of study until removal from treatment.
Time Frame: <1 cycle to 6 cycles of treatment
Measure: Median (Full Range); unit: months
Arm/Group | Oxaliplatin + Docetaxel
Number analyzed (Participants) | 15
months | 2.4 [0 to 6]

3. Secondary Outcome: Duration of Response
Description: Duration of response is a measure of how long the participants response to therapy was maintained.
Time Frame: 0 -12 months
Measure: Median (Full Range); unit: months
Arm/Group | Oxaliplatin + Docetaxel
Number analyzed (Participants) | 15
months | 7.9 [0 to 12]

4. Secondary Outcome: Safety Objective is to Describe the Safety Profile of 1st Line Treatment by Recording Grade 3 and 4 Adverse Events Experienced by Participants in This Trial.
Description: Toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE V 3.0) and the incidence of any Grade 3 or 4 toxicities will be analyzed. Toxicity is assessed every cycle.
Time Frame: day one of cycle one until participant removed from trial
Population: all participants had adverse events
Measure: Number; unit: participants
Arm/Group | Oxaliplatin + Docetaxel
Number analyzed (Participants) | 15
participants
  Grade 3 or 4 anemia | 1
  grade 3 or 4 thrombocytopenia | 1
  Grade 3 or 4 fatigue | 5
  Grade 3 or 4 dehydration | 2
  Grade 3 or 4 nausea | 1
  Grade 3 or 4 diarrhea | 2
  Grade 3 or 4 anorexia | 1
  Grade 3 or 4 neutropenia | 3
  Grade 3 or 4 vomiting | 2

ADVERSE EVENTS:
Arm/Group | Oxaliplatin + Docetaxel
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin + Docetaxel (N=15)
Catheter infection (Infections and infestations) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1)
clostridium difficile colitis (Gastrointestinal disorders) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
pain (Nervous system disorders) | 1 (1)
chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pericardial effusion (Cardiac disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DVT (Blood and lymphatic system disorders) | 1 (1)
concussion (Injury, poisoning and procedural complications) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin + Docetaxel (N=15)
Headache (Nervous system disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 10 (10)
vomiting (Gastrointestinal disorders) | 2 (2)
fatigue (General disorders) | 7 (7)
anorexia (Metabolism and nutrition disorders) | 3 (3)
dehydration (Metabolism and nutrition disorders) | 3 (3)
dysguesia (Nervous system disorders) | 5 (5)
alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
diarrhea (Gastrointestinal disorders) | 6 (6)
constipation (Gastrointestinal disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
neuropathy (Nervous system disorders) | 12 (12)
anemia (Blood and lymphatic system disorders) | 12 (12)
thrombocytopenia (Vascular disorders) | 5 (5)
neutropenia (Blood and lymphatic system disorders) | 6 (6)

LIMITATIONS AND CAVEATS:
Due to lack of recruitment, the study was closed early and conclusions should not necessarily be drawn from the data presented for duration of response

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes